CLINICAL TRIAL: NCT00397124
Title: Does the Vagus Nerve Play a Role in Tumor-to-Brain Communication? a Preliminary Study in Patients With Newly Diagnosed Lung Cancer
Brief Title: The Role of the Vagus Nerve in Tumor-to-Brain Communication in Lung Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: vagusCTIL
Record Dates: First submitted 2006-11-07; First posted 2006-11-08 (Estimated); Last update posted 2006-11-08 (Estimated); Status verified 2006-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

INTERVENTIONS:
Device: PET/CT imaging

SUMMARY:
the aim of this study is to measure brain metabolism in patients with lung cancer.FDG uptake in the brain in patients with malignant tumors will be compared to the amount of tracer activity found in patients who have benign pulmonary process. if differences between the brain uptake of FDG in the two groups will be found, further assessment will be performed in order to evaluate if such differences could be attributed and specifically localized to the brain regions innervated by the vagus

ELIGIBILITY:
Inclusion Criteria:

* patients with SPN referred for routine whole body FDG-PET imaging
* patients with NSCLC and patients with no evidence of lung cancer on further follow up

Exclusion Criteria:

* patients with a clinical history of vagotomy, abdominal surgery. brain tumor, brain trauma or CVA. or those with a systemic inflammatory disease

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-04

PRIMARY OUTCOMES:
the impact of the imaging modality on patients management

SECONDARY OUTCOMES:
the impact of the imaging modality on patients management

CONTACTS AND LOCATIONS:
Overall Officials: Ora Israel, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel